CLINICAL TRIAL: NCT02224898
Title: Feasibility of a Mobile Electronic Mindfulness Therapy Service for Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Walter G. Park, M.D., M.S., Principal Investigator, Stanford University
Other Study IDs: IRB-30976
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Pancreatitis, Chronic
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Definite/Suspected Chronic Pancreatitis: Patients with diagnosis of chronic pancreatitis with at least two of the following features: clinical course consistent with chronic pancreatitis, calcification in the pancreas on US/CT/EUS, ERCP showing ductal abnormalities (Cambridge Classification), exocrine insufficiency, histology showing irregular fibrosis, acinar cell loss, islet cell loss, and inflammatory cell infiltrates, or other features suggestive of chronic pancreatitis (such as pancreatic pseudocyst). The study group will also include patients with suspected chronic pancreatitis based on history of documented pancreatitis with lingering symptoms or signs of early chronic pancreatitis on imaging. Subjects will be asked to complete 30 days of mobile mindfulness therapy, for 2-30 minutes daily.
  Interventions: Behavioral: Mobile Mindfulness Therapy
- Healthy Control Group: Patients with no history of chronic gastrointestinal symptoms lasting greater than 8 weeks, no gastrointestinal disease or condition diagnosis, and are not currently experiencing gastrointestinal symptoms. Subjects will be asked to complete 30 days of mobile mindfulness therapy, for 2-30 minutes daily.
  Interventions: Behavioral: Mobile Mindfulness Therapy

INTERVENTIONS:
Behavioral: Mobile Mindfulness Therapy — Subjects will be asked to complete 30 days of mobile mindfulness therapy, for 2-30 minutes daily.

SUMMARY:
The research objective of this pilot study is to test the feasibility of a mobile electronic mindfulness therapy service for patients with definite or suspected chronic pancreatitis.

A secondary aim will be to determine the effect of the intervention on a symptom severity/global assessment of improvement for patients with chronic pancreatitis. The investigators hypothesize that a one-month period of daily mindfulness therapy delivered via a phone messaging service will reduce symptoms.

DETAILED DESCRIPTION:
Patients who meet diagnostic criteria for definite or suspected chronic pancreatitis and have current symptoms over the past month will be considered for study enrollment. Potential patients will be initially pre-screened by a patient chart review.

If not excluded during the pre-screening process, potential subjects will be mailed questionnaires to fill out at home and speak with a member of the research team for an intake interview. At that time, they will be asked to sign a consent form after its review. Subjects will then be given instructions on how to participate in daily mindfulness therapy for one-month via the phone messaging service with a research team member.

The total duration of the study intervention will be four weeks where enrolled patients will be asked to perform daily mindfulness sessions through our electronic mobile mindfulness therapy service.

Patients will be sent a daily automated text message or call reminder to their mobile phone at a pre-determined time, selected by the patient at the intake interview. The text message will prompt patients with a phone number to call to access the Mindfulness Therapy sessions.

When the patient is ready, s/he will call the provided phone number which is an automated answering and voice messaging service, which will prompt the patient to select a mindfulness therapy session of varying durations from 2 to 30 minutes. The session will lead the patients through deep relaxation breathing exercise for the duration the patient selected from the phone menu. Although the investigators will only ask patients to do one mindfulness session a day, patients are free to do as many as they want a day. At the end of their session, patients will leave a voice message with their name and current location such as home or work. The investigators will track the mindfulness sessions the individual patient participated in by obtaining their recorded voice messages in an inbox that correlates with the duration of the mindfulness session that the patient participated in. The voice messaging system will also provide information of the time the voice message was left, or time of completion of the patient's mindfulness session. If the patient prematurely terminated his/her session, got disconnected from his/her session or forgot to leave a message, the patient may call the same provided phone number to leave a message with his/her name, date of unrecorded session along with its duration and location of participation such as home or work.

At the end of the study at four weeks, patients will be asked to complete an exit interview. The patient will be asked to fill out questionnaires during this interview. The patient will also be asked to participate in an informal exit interview with one of the research team members. Patients will be asked of any new medications were added during the duration of the study. They will also be asked regarding any changes in chronic pancreatitis strategies and any new stressors.

ELIGIBILITY:
Inclusion Criteria:

* For the study group: Patients with diagnosis of chronic pancreatitis with at least two of the following features: clinical course consistent with chronic pancreatitis, calcification in the pancreas on US/CT/EUS, ERCP showing ductal abnormalities (Cambridge Classification), exocrine insufficiency, histology showing irregular fibrosis, acinar cell loss, islet cell loss, and inflammatory cell infiltrates, or other features suggestive of chronic pancreatitis (such as pancreatic pseudocyst). The study group will also include patients with suspected chronic pancreatitis based on history of documented pancreatitis with lingering symptoms or signs of early chronic pancreatitis on imaging.
* For the control group: no history of chronic GI symptoms lasting greater than 8 weeks, no gastrointestinal disease or condition diagnosis, and not be currently experiencing gastrointestinal symptoms.
* Age 18 to 80
* Willing to give informed consent
* Able to complete entire study
* Ability to speak and read English
* Regular menstrual cycles or menopause for at least 6 months
* Owns a mobile phone with texting capabilities
* Unlimited minutes and text messaging dataplan for mobile phone
* Physically and mentally capable of using a mobile phone
* Phone access

Exclusion Criteria:

* Red flags of concern: anemia, blood in stools, unexplained weight loss, unexplained fevers
* Pregnant or nursing woman, or planning on becoming pregnant within next year
* Travel plans outside of the county over the study duration or a month prior
* Change in medications one month prior or during study
* Change in chronic pancreatitis management strategies one month prior or during study such as dietary changes, exercise, counseling and behavioral therapies.
* Current co-morbid condition that might account for GI symptoms
* Current infectious diseases: HIV, Hepatitis A, B or C, other
* Psychiatric Conditions: moderate to severe depression (ECT, unable to work, disrupts ADL's), moderate to severe anxiety (unable to work, disrupts ADL's), bipolar disorder, schizophrenia, or history of psychosis, suicidal ideation or attempt, substance abuse (alcohol and/or drugs in past year), dissociative disorder, dementia related disorder
* Immunologic Diseases: systemic lupus, moderate to severe arthritis, scleroderma, other
* Gastrointestinal Disorders: inflammatory bowel diseases (ulcerative colitis, Crohn's), celiac disease,personal history of colon cancer or polyps, other unless condition associated with chronic pancreatitis.
* Cardiovascular disorder, clinically significant in past 12 months
* Pain disorder, clinically significant (back pain, fibromyalgia)
* Recent surgery, during 6 months prior to study enrollment or during study period (except minor surgeries such as wisdom teeth extraction, cataract surgery, corrective lens surgery, and/or minor skin surgeries)
* Major stressor(s) in life 3 months prior to study or anticipated over the next month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit a minimum of 10 and maximum of 40 subjects diagnosed with chronic pancreatitis and 5 healthy control subjects with no past or present chronic gastrointestinal symptoms lasting greater than 8 weeks, no chronic medical conditions and no organic gastrointestinal disease. All patients with suspected/definite chronic pancreatitis will be associated with Stanford Hospital and Clinics and the 5 healthy controls may or may not be associated with Stanford.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of a Mobile Mindfulness Therapy Application for Chronic Pancreatitis | 1 month
  The primary outcome will measure daily compliance rates with the denominator being 30 days and the numerator equal to the number of days out of 30 that the patient used the mobile mindfulness therapy application.

SECONDARY OUTCOMES:
The effect of mobile mindfulness therapy on a symptom severity/global assessment of improvement for patients with definite or suspected chronic pancreatitis | 1 month
  After consent to participate, the patient will complete a set of quality of life instruments before participating in the mindfulness therapy sessions. After 30 days, the patient will repeat completing the set of quality of life instruments. These include the SF-36, PANQOLI, and specific PROMIS QoL instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Park, MD, Principal Investigator — Stanford Hospital
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States